CLINICAL TRIAL: NCT04466670
Title: Dynamics of Hemostatic Parameters in COVID-19 and Comparison of Intervention Strategies Through Adaptive Clinical Trial
Brief Title: Hemostasis in COVID-19: an Adaptive Clinical Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Vanderson Geraldo Rocha, Full professor, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 33788820.9.0000.0068
Record Dates: First submitted 2020-07-08; First posted 2020-07-10 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; Thrombosis; Coagulopathy; Anticoagulation; Respiratory failure
MeSH Terms: conditions — COVID-19; Thrombosis; Hemostatic Disorders; Respiratory Insufficiency | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- phase 1 (No Intervention): Observational arm
- phase 2A (Experimental): Acetylsalicylic acid
  Interventions: Drug: acetylsalicylic acid
- phase 2B (Experimental): inhaled unfractionated heparin
  Interventions: Drug: Unfractionated heparin nebulized
- Placebo (Placebo Comparator): Placebo arm for Phase 2A
  Interventions: Drug: acetylsalicylic acid

INTERVENTIONS:
Drug: acetylsalicylic acid — acetylsalicylic acid (ASA) 100 mg daily PO up to 14 days OR arterial oxygen saturation greater than or equal to 92% on room air OR PaO2 to FiO2 ratio greater than 200 for 2 consecutive days, whichever is first.
  Other Names: aspirin
  Arms: Placebo; phase 2A
Drug: Unfractionated heparin nebulized — unfractionated heparin - 25,000 U/ 5 ml nebulized inhalation every 6 hours up to 14 days OR arterial oxygen saturation greater than or equal to 92% on room air OR PaO2 to FiO2 ratio greater than 200 for 2 consecutive days, whichever is first.
  Arms: phase 2B

SUMMARY:
Hypercoagulability has been demonstrated in COVID-19, leading to respiratory distress and increased mortality. This is an adaptive clinical trial to compare the efficacy and safety of two experimental strategies in patients with COVID-19: ASA or inhaled UFH associated with standard VTE prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥18 years of age at time of enrollment
* Subjects with a positive COVID-19 diagnosis by RT-PCR or serologic testing
* Subject (or legally authorized representative) must be willing, understanding and able to provide written informed consent.
* Only at phase 2:

  * onset of symptoms must not exceed 4 weeks
  * ICU patients
  * PaO2 to FiO2 ratio < 200

Exclusion Criteria:

1. General

   * Indications for therapeutic anticoagulation
   * History of chronic lung disease oxygen dependent
   * Pregnancy
   * Death considered imminent and inevitable within 24 hours
   * Patients under exclusive palliative care
   * Participation in another trial of investigational drug
   * Body weight < 40 Kg
   * Total bilirubin > 20 mg/dL
   * Severe active bleeding
   * Persistent GI bleeding
   * Known allergy to UFH or LMWH
   * History of heparin-induced thrombocytopenia (HIT) within the past 6 months
2. Exclusion criteria at phase 1

   * Platelet count < 25,000/mm3
   * Bacterial endocarditis
3. Exclusion criteria at phase 2

   * Platelet count < 50,000/mm3
   * History of surgery in the last 30 days
   * Intervention A: allergy to ASA and long-term use of antiplatelet drug
   * Intervention B: inhaled nitric oxide use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 379 (Estimated)
Dates: Start 2020-07-11 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Hospital discharge - alive / death | 30 days
  Number of COVID-19 positive patients who are alive within 30 days of symptoms onset

SECONDARY OUTCOMES:
Length of mechanical ventilation free days | 30 days
  Comparison of length of mechanical ventilation free days between each treatment arm
Length of renal replacement therapy free days | 30 days
  Comparison of length of renal replacement therapy free days between each treatment arm
Number of documented venous thromboembolism or arterial thrombosis | 3 months
  Comparison of number of thrombosis events between each treatment arm.

CONTACTS AND LOCATIONS:
Overall Officials: Vanderson Rocha, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- Vanderson Rocha, São Paulo, Brazil

REFERENCES:
- [Background] Schulman S, Kearon C; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in non-surgical patients. J Thromb Haemost. 2005 Apr;3(4):692-4. doi: 10.1111/j.1538-7836.2005.01204.x. PMID 15842354
- [Result] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Result] Fu L, Wang B, Yuan T, Chen X, Ao Y, Fitzpatrick T, Li P, Zhou Y, Lin YF, Duan Q, Luo G, Fan S, Lu Y, Feng A, Zhan Y, Liang B, Cai W, Zhang L, Du X, Li L, Shu Y, Zou H. Clinical characteristics of coronavirus disease 2019 (COVID-19) in China: A systematic review and meta-analysis. J Infect. 2020 Jun;80(6):656-665. doi: 10.1016/j.jinf.2020.03.041. Epub 2020 Apr 10. PMID 32283155
- [Result] Arachchillage DRJ, Laffan M. Abnormal coagulation parameters are associated with poor prognosis in patients with novel coronavirus pneumonia. J Thromb Haemost. 2020 May;18(5):1233-1234. doi: 10.1111/jth.14820. No abstract available. PMID 32291954
- [Result] Lillicrap D. Disseminated intravascular coagulation in patients with 2019-nCoV pneumonia. J Thromb Haemost. 2020 Apr;18(4):786-787. doi: 10.1111/jth.14781. Epub 2020 Mar 24. No abstract available. PMID 32212240
- [Result] Lippi G, Favaloro EJ. D-dimer is Associated with Severity of Coronavirus Disease 2019: A Pooled Analysis. Thromb Haemost. 2020 May;120(5):876-878. doi: 10.1055/s-0040-1709650. Epub 2020 Apr 3. No abstract available. PMID 32246450
- [Result] Feng Y, Ling Y, Bai T, Xie Y, Huang J, Li J, Xiong W, Yang D, Chen R, Lu F, Lu Y, Liu X, Chen Y, Li X, Li Y, Summah HD, Lin H, Yan J, Zhou M, Lu H, Qu J. COVID-19 with Different Severities: A Multicenter Study of Clinical Features. Am J Respir Crit Care Med. 2020 Jun 1;201(11):1380-1388. doi: 10.1164/rccm.202002-0445OC. PMID 32275452
- [Result] Cui S, Chen S, Li X, Liu S, Wang F. Prevalence of venous thromboembolism in patients with severe novel coronavirus pneumonia. J Thromb Haemost. 2020 Jun;18(6):1421-1424. doi: 10.1111/jth.14830. Epub 2020 May 6. PMID 32271988
- [Result] Klok FA, Kruip MJHA, van der Meer NJM, Arbous MS, Gommers DAMPJ, Kant KM, Kaptein FHJ, van Paassen J, Stals MAM, Huisman MV, Endeman H. Incidence of thrombotic complications in critically ill ICU patients with COVID-19. Thromb Res. 2020 Jul;191:145-147. doi: 10.1016/j.thromres.2020.04.013. Epub 2020 Apr 10. PMID 32291094
- [Result] Helms J, Tacquard C, Severac F, Leonard-Lorant I, Ohana M, Delabranche X, Merdji H, Clere-Jehl R, Schenck M, Fagot Gandet F, Fafi-Kremer S, Castelain V, Schneider F, Grunebaum L, Angles-Cano E, Sattler L, Mertes PM, Meziani F; CRICS TRIGGERSEP Group (Clinical Research in Intensive Care and Sepsis Trial Group for Global Evaluation and Research in Sepsis). High risk of thrombosis in patients with severe SARS-CoV-2 infection: a multicenter prospective cohort study. Intensive Care Med. 2020 Jun;46(6):1089-1098. doi: 10.1007/s00134-020-06062-x. Epub 2020 May 4. PMID 32367170
- [Result] Lodigiani C, Iapichino G, Carenzo L, Cecconi M, Ferrazzi P, Sebastian T, Kucher N, Studt JD, Sacco C, Bertuzzi A, Sandri MT, Barco S; Humanitas COVID-19 Task Force. Venous and arterial thromboembolic complications in COVID-19 patients admitted to an academic hospital in Milan, Italy. Thromb Res. 2020 Jul;191:9-14. doi: 10.1016/j.thromres.2020.04.024. Epub 2020 Apr 23. PMID 32353746
- [Result] Middeldorp S, Coppens M, van Haaps TF, Foppen M, Vlaar AP, Muller MCA, Bouman CCS, Beenen LFM, Kootte RS, Heijmans J, Smits LP, Bonta PI, van Es N. Incidence of venous thromboembolism in hospitalized patients with COVID-19. J Thromb Haemost. 2020 Aug;18(8):1995-2002. doi: 10.1111/jth.14888. Epub 2020 Jul 27. PMID 32369666
- [Result] Llitjos JF, Leclerc M, Chochois C, Monsallier JM, Ramakers M, Auvray M, Merouani K. High incidence of venous thromboembolic events in anticoagulated severe COVID-19 patients. J Thromb Haemost. 2020 Jul;18(7):1743-1746. doi: 10.1111/jth.14869. Epub 2020 May 27. PMID 32320517
- [Result] Gralinski LE, Bankhead A 3rd, Jeng S, Menachery VD, Proll S, Belisle SE, Matzke M, Webb-Robertson BJ, Luna ML, Shukla AK, Ferris MT, Bolles M, Chang J, Aicher L, Waters KM, Smith RD, Metz TO, Law GL, Katze MG, McWeeney S, Baric RS. Mechanisms of severe acute respiratory syndrome coronavirus-induced acute lung injury. mBio. 2013 Aug 6;4(4):e00271-13. doi: 10.1128/mBio.00271-13. PMID 23919993
- [Result] Walls AC, Park YJ, Tortorici MA, Wall A, McGuire AT, Veesler D. Structure, Function, and Antigenicity of the SARS-CoV-2 Spike Glycoprotein. Cell. 2020 Apr 16;181(2):281-292.e6. doi: 10.1016/j.cell.2020.02.058. Epub 2020 Mar 9. PMID 32155444
- [Result] Hoffmann M, Kleine-Weber H, Schroeder S, Kruger N, Herrler T, Erichsen S, Schiergens TS, Herrler G, Wu NH, Nitsche A, Muller MA, Drosten C, Pohlmann S. SARS-CoV-2 Cell Entry Depends on ACE2 and TMPRSS2 and Is Blocked by a Clinically Proven Protease Inhibitor. Cell. 2020 Apr 16;181(2):271-280.e8. doi: 10.1016/j.cell.2020.02.052. Epub 2020 Mar 5. PMID 32142651
- [Result] Hamming I, Timens W, Bulthuis ML, Lely AT, Navis G, van Goor H. Tissue distribution of ACE2 protein, the functional receptor for SARS coronavirus. A first step in understanding SARS pathogenesis. J Pathol. 2004 Jun;203(2):631-7. doi: 10.1002/path.1570. PMID 15141377
- [Result] Vaduganathan M, Vardeny O, Michel T, McMurray JJV, Pfeffer MA, Solomon SD. Renin-Angiotensin-Aldosterone System Inhibitors in Patients with Covid-19. N Engl J Med. 2020 Apr 23;382(17):1653-1659. doi: 10.1056/NEJMsr2005760. Epub 2020 Mar 30. No abstract available. PMID 32227760
- [Result] Ackermann M, Verleden SE, Kuehnel M, Haverich A, Welte T, Laenger F, Vanstapel A, Werlein C, Stark H, Tzankov A, Li WW, Li VW, Mentzer SJ, Jonigk D. Pulmonary Vascular Endothelialitis, Thrombosis, and Angiogenesis in Covid-19. N Engl J Med. 2020 Jul 9;383(2):120-128. doi: 10.1056/NEJMoa2015432. Epub 2020 May 21. PMID 32437596
- [Result] Dolhnikoff M, Duarte-Neto AN, de Almeida Monteiro RA, da Silva LFF, de Oliveira EP, Saldiva PHN, Mauad T, Negri EM. Pathological evidence of pulmonary thrombotic phenomena in severe COVID-19. J Thromb Haemost. 2020 Jun;18(6):1517-1519. doi: 10.1111/jth.14844. No abstract available. PMID 32294295
- [Result] Panigada M, Bottino N, Tagliabue P, Grasselli G, Novembrino C, Chantarangkul V, Pesenti A, Peyvandi F, Tripodi A. Hypercoagulability of COVID-19 patients in intensive care unit: A report of thromboelastography findings and other parameters of hemostasis. J Thromb Haemost. 2020 Jul;18(7):1738-1742. doi: 10.1111/jth.14850. Epub 2020 Jun 24. PMID 32302438
- [Result] Escher R, Breakey N, Lammle B. Severe COVID-19 infection associated with endothelial activation. Thromb Res. 2020 Jun;190:62. doi: 10.1016/j.thromres.2020.04.014. Epub 2020 Apr 15. No abstract available. PMID 32305740
- [Result] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578
- [Result] Whyte CS, Morrow GB, Mitchell JL, Chowdary P, Mutch NJ. Fibrinolytic abnormalities in acute respiratory distress syndrome (ARDS) and versatility of thrombolytic drugs to treat COVID-19. J Thromb Haemost. 2020 Jul;18(7):1548-1555. doi: 10.1111/jth.14872. Epub 2020 Jun 3. PMID 32329246
- [Result] White D, MacDonald S, Bull T, Hayman M, de Monteverde-Robb R, Sapsford D, Lavinio A, Varley J, Johnston A, Besser M, Thomas W. Heparin resistance in COVID-19 patients in the intensive care unit. J Thromb Thrombolysis. 2020 Aug;50(2):287-291. doi: 10.1007/s11239-020-02145-0. PMID 32445064
- [Result] Garcia DA, Baglin TP, Weitz JI, Samama MM. Parenteral anticoagulants: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e24S-e43S. doi: 10.1378/chest.11-2291. PMID 22315264
- [Result] Barrett CD, Moore HB, Yaffe MB, Moore EE. ISTH interim guidance on recognition and management of coagulopathy in COVID-19: A comment. J Thromb Haemost. 2020 Aug;18(8):2060-2063. doi: 10.1111/jth.14860. Epub 2020 Jun 14. No abstract available. PMID 32302462
- [Result] Bikdeli B, Madhavan MV, Jimenez D, Chuich T, Dreyfus I, Driggin E, Nigoghossian C, Ageno W, Madjid M, Guo Y, Tang LV, Hu Y, Giri J, Cushman M, Quere I, Dimakakos EP, Gibson CM, Lippi G, Favaloro EJ, Fareed J, Caprini JA, Tafur AJ, Burton JR, Francese DP, Wang EY, Falanga A, McLintock C, Hunt BJ, Spyropoulos AC, Barnes GD, Eikelboom JW, Weinberg I, Schulman S, Carrier M, Piazza G, Beckman JA, Steg PG, Stone GW, Rosenkranz S, Goldhaber SZ, Parikh SA, Monreal M, Krumholz HM, Konstantinides SV, Weitz JI, Lip GYH; Global COVID-19 Thrombosis Collaborative Group, Endorsed by the ISTH, NATF, ESVM, and the IUA, Supported by the ESC Working Group on Pulmonary Circulation and Right Ventricular Function. COVID-19 and Thrombotic or Thromboembolic Disease: Implications for Prevention, Antithrombotic Therapy, and Follow-Up: JACC State-of-the-Art Review. J Am Coll Cardiol. 2020 Jun 16;75(23):2950-2973. doi: 10.1016/j.jacc.2020.04.031. Epub 2020 Apr 17. PMID 32311448
- [Result] Maatman TK, Jalali F, Feizpour C, Douglas A 2nd, McGuire SP, Kinnaman G, Hartwell JL, Maatman BT, Kreutz RP, Kapoor R, Rahman O, Zyromski NJ, Meagher AD. Routine Venous Thromboembolism Prophylaxis May Be Inadequate in the Hypercoagulable State of Severe Coronavirus Disease 2019. Crit Care Med. 2020 Sep;48(9):e783-e790. doi: 10.1097/CCM.0000000000004466. PMID 32459672
- [Result] Nahum J, Morichau-Beauchant T, Daviaud F, Echegut P, Fichet J, Maillet JM, Thierry S. Venous Thrombosis Among Critically Ill Patients With Coronavirus Disease 2019 (COVID-19). JAMA Netw Open. 2020 May 1;3(5):e2010478. doi: 10.1001/jamanetworkopen.2020.10478. PMID 32469410
- [Result] Tremblay D, van Gerwen M, Alsen M, Thibaud S, Kessler A, Venugopal S, Makki I, Qin Q, Dharmapuri S, Jun T, Bhalla S, Berwick S, Feld J, Mascarenhas J, Troy K, Cromwell C, Dunn A, Oh WK, Naymagon L. Impact of anticoagulation prior to COVID-19 infection: a propensity score-matched cohort study. Blood. 2020 Jul 2;136(1):144-147. doi: 10.1182/blood.2020006941. No abstract available. PMID 32462179
- [Result] Paranjpe I, Fuster V, Lala A, Russak AJ, Glicksberg BS, Levin MA, Charney AW, Narula J, Fayad ZA, Bagiella E, Zhao S, Nadkarni GN. Association of Treatment Dose Anticoagulation With In-Hospital Survival Among Hospitalized Patients With COVID-19. J Am Coll Cardiol. 2020 Jul 7;76(1):122-124. doi: 10.1016/j.jacc.2020.05.001. Epub 2020 May 6. No abstract available. PMID 32387623
- [Result] Juschten J, Tuinman PR, Juffermans NP, Dixon B, Levi M, Schultz MJ. Nebulized anticoagulants in lung injury in critically ill patients-an updated systematic review of preclinical and clinical studies. Ann Transl Med. 2017 Nov;5(22):444. doi: 10.21037/atm.2017.08.23. PMID 29264361
- [Result] Dixon B, Schultz MJ, Smith R, Fink JB, Santamaria JD, Campbell DJ. Nebulized heparin is associated with fewer days of mechanical ventilation in critically ill patients: a randomized controlled trial. Crit Care. 2010;14(5):R180. doi: 10.1186/cc9286. Epub 2010 Oct 11. PMID 20937093
- [Result] Viecca M, Radovanovic D, Forleo GB, Santus P. Enhanced platelet inhibition treatment improves hypoxemia in patients with severe Covid-19 and hypercoagulability. A case control, proof of concept study. Pharmacol Res. 2020 Aug;158:104950. doi: 10.1016/j.phrs.2020.104950. Epub 2020 May 23. PMID 32450344
- [Result] Connor JT, Elm JJ, Broglio KR; ESETT and ADAPT-IT Investigators. Bayesian adaptive trials offer advantages in comparative effectiveness trials: an example in status epilepticus. J Clin Epidemiol. 2013 Aug;66(8 Suppl):S130-7. doi: 10.1016/j.jclinepi.2013.02.015. PMID 23849147
- [Result] Gsponer T, Gerber F, Bornkamp B, Ohlssen D, Vandemeulebroecke M, Schmidli H. A practical guide to Bayesian group sequential designs. Pharm Stat. 2014 Jan-Feb;13(1):71-80. doi: 10.1002/pst.1593. Epub 2013 Aug 24. PMID 24038922